CLINICAL TRIAL: NCT05863208
Title: Comparison of The Adenoma Detection Rate Between Artificial Intelligence-assisted Colonoscopy With or Without Endocuff Vision and Standard Colonscopy: A Randomized Controlled Study
Brief Title: Artificial Intelligence-assisted Colonoscopy With or Without Endocuff Vision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EMRP53109N
Record Dates: First submitted 2023-05-09; First posted 2023-05-17 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Adenoma Detection Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Artificial Intelligence-assisted Colonoscopy with Endocuff Vision (Active Comparator): Use artificial intelligence-assisted colonoscopy with Endocuff Vision
  Interventions: Device: Artificial intelligence; Device: Endocuff vision; Device: High-definition endoscope
- Artificial Intelligence-assisted Colonoscopy (Active Comparator): Use artificial intelligence-assisted colonoscopy alone
  Interventions: Device: Artificial intelligence; Device: High-definition endoscope
- Standard colonoscopy (Sham Comparator): Use standard colonoscopy without artificial intelligence-assisted colonoscopy or Endocuff Vision
  Interventions: Device: High-definition endoscope

INTERVENTIONS:
Device: Artificial intelligence — ASUS EndoAim AI Endoscopy System (ASUS, Taiwan) is used to help the detection of colon adenoma
  Arms: Artificial Intelligence-assisted Colonoscopy; Artificial Intelligence-assisted Colonoscopy with Endocuff Vision
Device: Endocuff vision — Endocuff vision (Olympus, UK) is used to help the detection of colon adenoma
  Arms: Artificial Intelligence-assisted Colonoscopy with Endocuff Vision
Device: High-definition endoscope — High-definition endoscope (EVIS-EXERA 290 video system, Olympus Optical, Aizu, Japan) is used under white light for the detection of colon adenoma

SUMMARY:
Adenoma detection rate (ADR) is considered the single most important quality measure in colonoscopy and a higher ADR can reduce the risk of interval colorectal cancer (CRC). Several kinds of new endoscopes and accessories have been accessed to investigate the abilities of improving the ADR. Artificial intelligence (AI) and Endocuff vision are promising new devices to improve the ADR. However, the effect of combining AI and Endocuff vision on ADR remains unclear. The aim of this prospective randomized study is to compare the ADR of AI plus Endocuff vision, AI alone and standard colonoscopy examination.

DETAILED DESCRIPTION:
This is a prospective single-blinded randomized controlled trial of three different types of colonoscopy examinations by 1:1:1 ratio. We use EndoAim AI (ASUS, Taiwan) and Endocuff vision (Olympus, UK) assisted colonoscopy in the first group. We use AI assisted colonoscopy in the 2nd group. We use standard colonoscopy in the 3rd group.

Eligible patients are older than 40 years old and receive colonoscopy for either symptomatic or screening/surveillance. All endoscopists should receive training on EndoAim AI systems and Endocuff vision. During the procedure, experienced endoscopists use high-definition endoscopes (EVIS-EXERA 290 video system, Olympus Optical, Aizu, Japan) under white light and insert to the cecum in the three different groups. The cecal intubation is confirmed by the identification of ileocecal valve and appendiceal orifice.

The Boston Bowel Preparation Scale is used for grading the bowel preparation quality. The size (compared with biopsy forceps), location and morphology of polyps are recorded by the independent endoscopist. All polyps ae removed by either biopsy or polypectomy. The insertion and withdrawal time are measured. The time of the polypectomy site is not included in the withdrawal time.

ELIGIBILITY:
Inclusion Criteria:

Patients over 20 years old are undergoing outpatient sedative colonoscopy in the E-Da Hospital, E-Da cancer Hospital and Chung Shan Medical University Hospital in Taiwan

Exclusion Criteria:

* A prior history of of inflammatory bowel disease, colorectal cancer, previous bowel resection, Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes
* Bleeding tendency
* For scheduled endoscopic treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | One month after colonoscopy
  The proportion of patients with at least one adenomas

SECONDARY OUTCOMES:
Polyp detection rate | One month after colonoscopy
  The proportion of patients with at least one polyp
Sessile serrated adenoma detection rate | One month after colonoscopy
  The proportion of patients with at least one sessile serrated adenoma
Sessile serrated polyps detection rate | One month after colonoscopy
  The proportion of patients with at least one sessile serrated polyp
Advanced adenoma detection rate | One month after colonoscopy
  The proportion of patients with at least one advanced adenoma
Mean number of polyp per patient | One month after colonoscopy
  The mean number of polyp per patient
Mean number of adenoma per patient | One month after colonoscopy
  The mean number of adenoma per patient
Total number of polyp or adenoma per patient | One month after colonoscopy
  The total number of polyp or adenoma per patient

CONTACTS AND LOCATIONS:
Overall Officials: Ying Nan Tsai, MD, Study Chair — Division of Gastroenterology and Hepatology, E-Da Cancer Hospital, Kaohsiung, Taiwan
Locations (1):
- E-DA Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Fernandez C, Garcia-Rangel D, Aguilar-Olivos NE, Barreto-Zuniga R, Romano-Munive AF, Grajales-Figueroa G, Zamora-Nava LE, Tellez-Avila FI. Higher adenoma detection rate with the endocuff: a randomized trial. Endoscopy. 2017 Nov;49(11):1061-1068. doi: 10.1055/s-0043-117879. Epub 2017 Sep 12. PMID 28898920
- [Background] Triantafyllou K, Polymeros D, Apostolopoulos P, Lopes Brandao C, Gkolfakis P, Repici A, Papanikolaou IS, Dinis-Ribeiro M, Alexandrakis G, Hassan C. Endocuff-assisted colonoscopy is associated with a lower adenoma miss rate: a multicenter randomized tandem study. Endoscopy. 2017 Nov;49(11):1051-1060. doi: 10.1055/s-0043-114412. Epub 2017 Aug 1. PMID 28763808
- [Background] Williet N, Tournier Q, Vernet C, Dumas O, Rinaldi L, Roblin X, Phelip JM, Pioche M. Effect of Endocuff-assisted colonoscopy on adenoma detection rate: meta-analysis of randomized controlled trials. Endoscopy. 2018 Sep;50(9):846-860. doi: 10.1055/a-0577-3500. Epub 2018 Apr 26. PMID 29698990
- [Background] Xu H, Tang RSY, Lam TYT, Zhao G, Lau JYW, Liu Y, Wu Q, Rong L, Xu W, Li X, Wong SH, Cai S, Wang J, Liu G, Ma T, Liang X, Mak JWY, Xu H, Yuan P, Cao T, Li F, Ye Z, Shutian Z, Sung JJY. Artificial Intelligence-Assisted Colonoscopy for Colorectal Cancer Screening: A Multicenter Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2023 Feb;21(2):337-346.e3. doi: 10.1016/j.cgh.2022.07.006. Epub 2022 Jul 19. PMID 35863686
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963